CLINICAL TRIAL: NCT03995641
Title: The Effect of Local Analgesia on Postoperative Gluteal Pain in Patients Undergoing Sacrospinous Ligament Fixation: A Randomized Trial
Brief Title: The Effect of Local Analgesia on Postoperative Gluteal Pain in Patients Undergoing Sacrospinous Ligament Fixation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Never received appropriate formulation.
Sponsor: Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-002
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Pain; Pelvic Organ Prolapse; Trigger Point Injection; Sacrospinous Ligament Fixation
MeSH Terms: conditions — Pain, Postoperative; Pelvic Organ Prolapse | interventions — Bupivacaine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery Alone (No Intervention): Patient will receive sacrospinous ligament suspension surgery without any additional interventions
- Surgery Plus Trigger Point Injection (Experimental): Patient will have sacrospinous ligament suspension procedure with addition of a trigger point injection (9cc of 0.5% marcaine and 1 cc kenalog) over area of suture placement
  Interventions: Drug: marcaine and kenalog

INTERVENTIONS:
Drug: marcaine and kenalog — Trigger point injection (consisting of 9 cc 0.5% Marcaine and 1 cc kenalog) may be given at time of surgery if patient is randomized to receive the injection
  Arms: Surgery Plus Trigger Point Injection

SUMMARY:
This study will randomize patients to either receive intraoperative administration of local anesthetic and corticosteriod at time of sacrospinous ligament fixation compared to placebo to determine if intraoperative trigger point injection (TPI) improves postoperative gluteal and sciatic pain scores along with use of narcotic pain medications.

There is a paucity of data examining interventions to potentially ameliorate the postoperative gluteal pain often associated with sacrospinous ligament colpopexy. Our study aims to determine if a compounded TPI improves postoperative pain scores and minimizes use of narcotic pain medications by 20% compared to controls.

DETAILED DESCRIPTION:
Sacrospinous ligament fixation (SSLF) is commonly performed to treat apical prolapse. Pelvic organ prolapse (POP) is a complaint for which as many as 11% of women seek surgical intervention in their lifetimes (2). SSLF is associated with shorter operating time, improved patient recovery time, fewer complications and decreased costs compared to an abdominal approach (3).This procedure is associated with postoperative nerve pain in 6.1% to 15.3% of SSLF procedures, due to impingement of the S3 to S5 nerve roots that course over the mid-portion of the coccygeus muscle-sacrospinous ligament (C-SSL) complex (1). 89% of the nerve fibers to the coccygeus and/or levator ani muscles (S3) course over the midportion of the C-SSL complex, just proximal to the intended location for suspension (4). This resulting nerve entrapment or injury may then lead to gluteal and perineal pain, parasthesias and muscle weakness (1). This pain may persist 6 weeks in up to 15% of patients,but most patients can be managed with conservative therapies, such as medications, TPIs and/or pelvic floor physical therapy (3).

A myofascial trigger point is a hyperirritable area in skeletal muscle that is painful on compression and can give rise to characteristic referred pain and tenderness, motor dysfunction and autonomic phenomena (5). TPIs are a treatment used in cases of chronic myofascial nerve pain and involve injection of the involved muscle(s), typically with local anesthetics and corticosteroids (5). The mechanism of action of TPIs occurs by mechanical disruption of abnormal contractile elements, dilution of nociceptive substances by the infiltrated anesthetic, and induction of muscle fiber trauma that subsequently releases intracellular potassium. Additionally, injections interrupt the positive feedback loop that perpetuates pain and a vasodilatory effect of anesthetic helps to remove excess metabolites (5). The benefits of this local combined pain control method are two-fold: the local anesthetic offers rapid pain relief for several hours while the corticosteroid provides delayed pain control, often lasting three to five weeks (6). The use of such local analgesia is not typically standard of care at the time of a sacrospinous ligament fixation, but may be a helpful adjunct therapy.

A recent case report noted significant improvement in a patient's pelvic pain after she received three therapeutic pudendal nerve perineal injections using the combination of a local anesthetic and steroid (bupivicaine 0.25% and triamcinolone 40 mg); two injections were placed at the ischial spine and one in Alcock's canal (7). Similarly, another randomized controlled trial found that injection of slow-release corticosteroid (triamcinolone) and lidocaine in the anatomic region around the sacrospinous ligament's insertion on the ischial spine (i.e., also in the area of SSL colpopexy) significantly reduced pain intensity and number of pain locations in women with persistent, debilitating sacral low back pain, even spanning up to two years after pregnancy and childbirth (8).

There is a paucity of data examining interventions to potentially ameliorate the postoperative transient gluteal pain often associated with sacrospinous ligament colpopexy. The only comparable study to date examined the injection of 0.25% bupivicaine at the time of sacrospinous ligament colpopexy and found that such an intervention did not reduce patient's perceptions of postoperative gluteal pain, but did potentially reduce the need for medication after surgery (1). Our study aims to determine if a compounded TPI (9cc 0.5% marcaine and 1cc Kenalog) improves postoperative gluteal pain scores and minimizes use of narcotic pain medications in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* 21yo or older
* English speaking
* Stage II or greater pelvic organ prolapse
* Sacrospinous Ligament Fixation (SSLF) used as apical suspension
* SSLF scheduled to be performed by Dr. Janelle Evans or Dr. Marc Ashby

Exclusion Criteria:

* Under 21yo
* Non English speaking
* Patient consented, but SSLF not performed at time of surgery
* Patient on chronic opiates preoperatively (greater than three months of use)
* Contraindication to Marcaine or Kenalog
* Prisoners and those involuntarily confined
* Patients with cognitive impairment or those using a legally-authorized representative
* Hysterectomy performed at time of suspension

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
objective pain score | 6 weeks postoperative
  morphine equivalents

SECONDARY OUTCOMES:
subjective pain score rating | 6 weeks postoperative
  pain scale 0-10 (no pain to severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Kettering Health Network, Dayton, Ohio, United States